CLINICAL TRIAL: NCT05475275
Title: A Prospective Randomized Controlled Trial of the Effect of Different Pancreaticojejunostomy After Pancreaticoduodenectomy on Postoperative Pancreatic Fistula Based on the Position of the Pancreatic Duct in Pancreatic Section
Brief Title: Different Pancreaticojejunostomy After Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Junjie Xiong (Other)
Responsible Party: Sponsor-Investigator, Junjie Xiong, associate chief physician, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022(148)
Record Dates: First submitted 2022-07-11; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Pancreaticoduodenectomy; Postoperative Pancreatic Fistula
Keywords: pancreaticoduodenectomy; pancreaticojejunostomy; postoperative pancreatic fistula; pancreatic duct
MeSH Terms: interventions — Pancreaticojejunostomy

STUDY DESIGN:
Intervention Model Description: The patients were randomly divided into the experimental group and the control group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Enclosed envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group underwent intraoperative measurements (A: short distance from the center of the pancreatic duct to the edge of the pancreas) and (B: pancreatic thickness). When the ratio of the thickness of the short distance from the center of the pancreatic duct to the edge of the pancreas at the pancreatic section was ≥0.401, it was divided into the N1 group (central pancreatic duct). If the ratio was <0.401, it was divided into the N2 group (eccentric pancreatic duct). The "central pancreatic duct" group was given "1+1 mode" pancreaticojejunostomy; the "eccentric pancreatic duct" group was given "1+1² mode" pancreaticojejunostomy.
  Interventions: Procedure: pancreaticojejunostomy
- Control group (Active Comparator): The patients in the control group were given "traditional pancreaticojejunostomy"
  Interventions: Procedure: pancreaticojejunostomy

INTERVENTIONS:
Procedure: pancreaticojejunostomy — The experimental group underwent intraoperative measurements (A: short distance from the center of the pancreatic duct to the edge of the pancreas) and (B: pancreatic thickness). When the ratio of the thickness of the short distance from the center of the pancreatic duct to the edge of the pancreas at the pancreatic section was ≥0.401, it was divided into the N1 group (central pancreatic duct). If the ratio was <0.401, it was divided into the N2 group (eccentric pancreatic duct). The "central pancreatic duct" group was given "1+1 mode" pancreaticojejunostomy; the "eccentric pancreatic duct" group was given "1+1² mode" pancreaticojejunostomy.

SUMMARY:
The aim of this study was to reduce the incidence of postoperative pancreatic fistula after pancreaticoduodenectomy by using different pancreaticojejunostomy methods according to the position of the pancreatic duct.

DETAILED DESCRIPTION:
Pancreatectomy, especially pancreaticoduodenectomy, is the most complicated surgical approach in all abdominal surgeries. Postoperative pancreatic fistula (POPF) is the most serious complication after pancreaticoduodenectomy. Once it occurs, it will affect postoperative recovery, increase abdominal infection, and even lead to postoperative hemorrhage and life-threatening conditions. The quality of pancreaticojejunostomy has an inevitable relationship with postoperative pancreatic fistula. At present, there are many studies based on the risk factors for pancreatic fistula, including the texture of the pancreas, the diameter of the pancreatic duct, the patient's general condition and other factors, but little attention has been given to the position of the pancreatic duct in the residual pancreatic section. At present, the choice of pancreaticojejunostomy is more arbitrary. Although duct-to-mucosa pancreaticojejunostomy has become mainstream, there are still great differences. At present, there is no pancreaticojejunostomy that can completely avoid the occurrence of pancreatic fistula. The investigators found that the anatomical position of the pancreatic duct in pancreatic section was very important in pancreaticoduodenectomy and divided them into the central type and eccentric type. It was initially found that the incidence of pancreatic fistula after an eccentric pancreatic duct was significantly increased. It was confirmed that the anatomical position of the pancreatic duct is related to the occurrence of POPF. On this basis, the investigators proposed that different types of pancreatic ducts using different anastomosis methods, which may reduce the incidence of POPF. The study data come from the Department of Pancreatic Surgery, West China Hospital, Sichuan University, and the sample size is estimated from the number of patients admitted to the Department of Pancreatic Surgery in the past two years according to the POPF rate. The participants were randomly divided into the experimental group and the control group. The experimental group underwent intraoperative measurements (A: short distance from the center of the pancreatic duct to the edge of the pancreas) and (B: pancreatic thickness). When the ratio of the thickness of the short distance from the center of the pancreatic duct to the edge of the pancreas at the pancreatic section was ≥0.401, it was divided into the N1 group (central pancreatic duct). If the ratio was <0.401, it was divided into the N2 group (eccentric pancreatic duct). The "central pancreatic duct" group was given "1+1 mode" pancreaticojejunostomy; the "eccentric pancreatic duct" group was given "1+1² mode" pancreaticojejunostomy. The patients in the control group were given "traditional pancreaticojejunostomy". The preoperative basic conditions and postoperative clinically relevant pancreatic fistula and other complications were compared between the two groups. This is expected to be confirmed by the investigators basing on the different types of pancreatic ducts, and the corresponding pancreaticojejunostomy can reduce the incidence of postoperative pancreatic fistula in patients undergoing pancreaticoduodenectomy. The primary outcome was the rate of POPF, and the secondary outcomes included postoperative hemorrhage, postoperative biliary fistula, delayed gastric emptying and so on. Preoperative baseline characteristic data were collected, including age, sex, BMI, ASA, preoperative serum protein level, preoperative blood total bilirubin level, and so on. The postoperative complications and recovery data were collected.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of benign or malignant peri-ampullary diseases
* The participants have age more than18 years
* The participants have adequate organ function to tolerate surgery

Exclusion Criteria:

*The participants undergoing other organ surgery at the same time

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 924 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula(POPF) as assessed by 2016 ISGPS definition | Within 30 days
  2016 ISGPS definition(POPF):A drain output of any measurable volume of fluid with an amylase level >3 times the upper limit of institutional normal serum amylase activity, associated with a clinically relevant development/condition related directly to the postoperative pancreatic fistula.

SECONDARY OUTCOMES:
Postoperative hemorrhage as assessed by ISGPS definition | Within 30 days
  Postoperative hemorrhage(ISGPS definition):definition of PPH is based on three parameters: time of onset, location, and severity of hemorrhage: (1)Onset is either early (≤24 hours after end of the index operation) or late (>24 hours); (2) Location is either intraluminal (eg,pancreatic surface, anastomoses, gastric/duodenal ulcer/erosion, or hemobilia) or extraluminal (eg, arterial or venous vessel, operating field, external suture or staple line, or pseudoaneurysm); (3) Severity of bleeding may be mild or severe.
Delayed gastric emptying as assessed by ISGPS definition | Within 30 days
  Delayed gastric emptying(ISGPS definition):Delayed gastric emptying represents the inability to return to a standard diet by the end of the first postoperative week and includes prolonged nasogastric intubation of the patient. Three different grades (A, B, and C) were defined based on the impact on the clinical course and on postoperative management.

CONTACTS AND LOCATIONS:
Overall Officials: Bole Tian, MD, Study Chair — West China Hospital
Locations (1):
- Bole Tian, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu C, Hou SZ, Wu Z, Huang X, Wang Z, Tian B. Prognostic Nomogram for patients undergoing radical Pancreaticoduodenectomy for adenocarcinoma of the pancreatic head. BMC Cancer. 2021 May 27;21(1):624. doi: 10.1186/s12885-021-08295-5. PMID 34044806
- [Result] Wang WG, Fu L, Babu SR, Wang L, Liang CP, Tian BL. Incidence of and Risk Factors and Reinterventions for Post-Pancreatoduodenectomy Hemorrhage: Retrospective Analysis. Dig Surg. 2018;35(1):19-27. doi: 10.1159/000460263. Epub 2017 Apr 7. PMID 28384642
- [Result] Su AP, Zhang Y, Ke NW, Lu HM, Tian BL, Hu WM, Zhang ZD. Triple-layer duct-to-mucosa pancreaticojejunostomy with resection of jejunal serosa decreased pancreatic fistula after pancreaticoduodenectomy. J Surg Res. 2014 Jan;186(1):184-91. doi: 10.1016/j.jss.2013.08.029. Epub 2013 Sep 21. PMID 24095023
- [Result] Su AP, Ke NW, Zhang Y, Wang WG, Zhang ZD, Liu XB, Hu WM, Tian BL. Does modified Braun enteroenterostomy improve alkaline reflux gastritis and marginal ulcer after pancreaticoduodenectomy? Dig Dis Sci. 2013 Nov;58(11):3224-31. doi: 10.1007/s10620-013-2803-x. Epub 2013 Aug 6. PMID 23918152
- [Result] Hirono S, Kawai M, Okada KI, Miyazawa M, Kitahata Y, Hayami S, Ueno M, Yamaue H. Modified Blumgart Mattress Suture Versus Conventional Interrupted Suture in Pancreaticojejunostomy During Pancreaticoduodenectomy: Randomized Controlled Trial. Ann Surg. 2019 Feb;269(2):243-251. doi: 10.1097/SLA.0000000000002802. PMID 29697455
- [Result] Ecker BL, McMillan MT, Asbun HJ, Ball CG, Bassi C, Beane JD, Behrman SW, Berger AC, Dickson EJ, Bloomston M, Callery MP, Christein JD, Dixon E, Drebin JA, Castillo CF, Fisher WE, Fong ZV, Haverick E, Hollis RH, House MG, Hughes SJ, Jamieson NB, Javed AA, Kent TS, Kowalsky SJ, Kunstman JW, Malleo G, Poruk KE, Salem RR, Schmidt CR, Soares K, Stauffer JA, Valero V, Velu LKP, Watkins AA, Wolfgang CL, Zureikat AH, Vollmer CM Jr. Characterization and Optimal Management of High-risk Pancreatic Anastomoses During Pancreatoduodenectomy. Ann Surg. 2018 Apr;267(4):608-616. doi: 10.1097/SLA.0000000000002327. PMID 28594741
- [Result] Keck T, Wellner UF, Bahra M, Klein F, Sick O, Niedergethmann M, Wilhelm TJ, Farkas SA, Borner T, Bruns C, Kleespies A, Kleeff J, Mihaljevic AL, Uhl W, Chromik A, Fendrich V, Heeger K, Padberg W, Hecker A, Neumann UP, Junge K, Kalff JC, Glowka TR, Werner J, Knebel P, Piso P, Mayr M, Izbicki J, Vashist Y, Bronsert P, Bruckner T, Limprecht R, Diener MK, Rossion I, Wegener I, Hopt UT. Pancreatogastrostomy Versus Pancreatojejunostomy for RECOnstruction After PANCreatoduodenectomy (RECOPANC, DRKS 00000767): Perioperative and Long-term Results of a Multicenter Randomized Controlled Trial. Ann Surg. 2016 Mar;263(3):440-9. doi: 10.1097/SLA.0000000000001240. PMID 26135690

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-07-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT05475275/SAP_000.pdf
  • Informed Consent Form (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT05475275/ICF_001.pdf